CLINICAL TRIAL: NCT07023211
Title: Neofunctional Deep Diaphragmatic Breathing Interventions for Stress Modulation: A Comparative RCT Assessing Physiological and Psychological Parameters
Brief Title: Neofunctional Deep Breathing for Stress Modulation
Acronym: SIRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Collaborators: Centro Studi Psicoterapia Neo-Funzionale (Unknown)
Responsible Party: Principal Investigator, Giuseppe Maniaci, Adjunct Professor, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOPalermo_2
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: diaphragmatic breathing; mind-body therapies; stress; vagal tone; social touch; Functional psychotherapy; parasympathetic nervous system

STUDY DESIGN:
Intervention Model Description: After a psychiatric, psychological and anthropometric assessment, healthy volunteers will receive the Trier Social Stress Test (TSST) procedure and then they are randomly assigned to 30 min of deep diaphragmatic breathing based on Functional Therapy (FT) or Social Touch (ST). All subjects are tested at the baseline (T0), at the end of the TSST (T1), and at the end of the treatment (T2).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects are advised that they are going to receive some kind of psychological support after a psychosocial stress. The investigator isn't informed about the randomisation procedures of the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Therapy (FT) (Experimental): Participants will be lying down in supine position. This breathing technique, rooted in the Neo-Functionalist orientation which actively utilizes body contact, involves direct manual assistance from the therapist during different respiratory movements. It is specifically aimed at promoting and facilitating congruent movements across the thoracic, diaphragmatic, and abdominal regions throughout the breathing cycle, enhancing the targeted respiratory pattern. The intervention will be delivered by a psychotherapist specialized in Neo-Functional techniques. Selected musical tracks accompany the session. The FT session will last 30 minutes.
  Interventions: Behavioral: Neo-Functional diaphragmatic breathing
- Social Touch (ST) (Sham Comparator): This group is designed to control for the variable of physical contact. Participants will receive occasional physical contact applied by the therapist specifically to the participant's right arm, while listening to the same musical tracks used in the experimental (FT) group. This contact is deliberately non-specific to the breathing process and contrasts with the targeted manual respiratory assistance provided to the experimental group. Participants in this group will not receive breathing instructions. The ST session will last 30 minutes.
  Interventions: Behavioral: Social touch

INTERVENTIONS:
Behavioral: Neo-Functional diaphragmatic breathing — This technique, rooted in the Neo-Functionalist orientation which actively utilizes body contact, involves direct manual assistance from the therapist during different respiratory movements. This hands-on guidance is specifically aimed at promoting and facilitating congruent movements across the thoracic, diaphragmatic, and abdominal regions throughout the breathing cycle, enhancing the targeted respiratory pattern. The intervention will be delivered by a psychotherapist specialized in Neo-Functional techniques.
  Arms: Functional Therapy (FT)
Behavioral: Social touch — Participants will receive occasional physical contact applied by the therapist specifically to the right arm. This contact is deliberately non-specific to the breathing process and contrasts with the targeted manual respiratory assistance provided to the experimental group. Participants in this group will not receive breathing instructions.
  Arms: Social Touch (ST)

SUMMARY:
The goal of this pilot randomized clinical trial is to learn if a single session of Neo-Functional diaphragmatic breathing can stimulate vagotonia and help to restore a state of relaxation after acute stress in healthy adult volunteers (male and female, aged 18-45). The main research question is: does a single 30-minute session of Neo-Functional diaphragmatic breathing intervention lead to better physiological (heart rate, skin conductance, muscle tension, abdominal excursion) and psychological (State-Trait Anxiety Inventory - State scale [STAI-State], Subjective Units of Distress Scale [SUDS]) recovery after an acute stressor (Trier Social Stress Test [TSST]) compared to a control condition? The study will compare an experimental group receiving the Neo-Functional diaphragmatic breathing intervention to a control group that rests in the presence of a therapist with minimal contact but without the specific breathing technique, to see if the breathing intervention results in a more significant reduction in stress markers and improvement in relaxation indicators. Participants will: undergo initial assessments including physiological measurements (heart rate [HR], skin conductance [SC], left deltoid surface electromyography [EMG], respiratory rate [breaths per minute, BPM] and respiratory amplitude [RESP AMP], derived from abdominal excursion), anthropometric measurements (weight, height, Body Mass Index [BMI]), and psychological questionnaires (STAI-State, SUDS); be subjected to the Trier Social Stress Test (TSST) to induce acute stress; undergo post-stress assessments (physiological and psychological); be randomly assigned to either receive a 30-minute Neo-Functional diaphragmatic breathing session (Experimental Group) or rest in the presence of a therapist (Control Group); undergo final physiological and psychological assessments.

DETAILED DESCRIPTION:
Modern life often exposes individuals to significant levels of stress, which can negatively impact both psychological well-being and physical health. Chronic stress is known to disrupt the body's natural balance, potentially affecting the immune system and contributing to various health problems. This interplay between the mind, nervous system, endocrine system, and immune system is studied within the field of Psycho-Neuro-Endocrino-Immunology (PNEI). Mind-Body Therapies (MBTs), such as Yoga, Mindfulness, and Qigong, often incorporate specific breathing techniques, particularly diaphragmatic breathing (deep, abdominal breathing), as a core component. These techniques are thought to exert their beneficial effects, at least in part, by stimulating the vagus nerve. The vagus nerve is a major component of the parasympathetic nervous system, often referred to as the "rest and digest" system, which counteracts the stress response ("fight or flight") driven by the sympathetic nervous system. Enhanced vagal tone is associated with better stress regulation, reduced inflammation, and improved overall health. This study focuses on a specific diaphragmatic breathing technique derived from the Neo-Functionalism theoretical orientation. This approach suggests that therapeutic interventions targeting bodily functions can influence psychological states. Uniquely, the Neo-Functional technique, as applied in this study, involves not only guided breathing instruction but also direct physical contact and specific breathing maneuvers. While the long-term benefits of various MBTs are increasingly documented, there is limited research, particularly using rigorous, controlled designs, investigating the immediate physiological and psychological effects of a single session of a specific, guided diaphragmatic breathing technique involving manual assistance following an acute stress exposure. Healthy volunteers will be recruited via advertisements. It is planned to enroll a sample of 40 participants (aged 18-45 years, balanced for sex). For initial screening, interested subjects will be evaluated by a psychologist or psychiatry resident using a structured diagnostic interview (Structured Clinical Interview for DSM-5 [SCID-5]) to exclude the presence of psychiatric disorders. All study assessments and procedures will take place at the premises of the Section of Psychiatry, Department of Biomedicine, Neurosciences and Advanced Diagnostics, at the "P. Giaccone" Polyclinic in Palermo. Following the initial assessment and confirmation of eligibility, subjects will be randomized to either the Experimental group or the Control group. All experimental sessions will occur in a controlled setting within the Section of Psychiatry. During the session, anthropometric, psychological, and physiological parameters via biofeedback will be assessed for each participant. Anthropometric parameters include height, weight, and Body Mass Index (BMI). Psychological assessment includes the State-Trait Anxiety Inventory (limited to the State scale - STAI-State) and the Subjective Units of Distress Scale (SUDS). Biofeedback parameters include heart rate (HR), skin conductance (SC), left deltoid surface electromyography (EMG), respiratory rate [breaths per minute, BPM] and respiratory amplitude [RESP AMP] derived from abdominal excursion, with biofeedback sensors remaining connected throughout the experimental procedure. Upon arrival (T0 - Baseline), anthropometric parameters will be assessed, then biofeedback sensors will be applied, and physiological parameters will be recorded at rest to establish the baseline; STAI-State and SUDS questionnaires will also be administered at this time. Subsequently, participants will undergo the Trier Social Stress Test (TSST), a standardized protocol used to induce psychophysiological stress under controlled conditions. The TSST is divided into 5-minute components and the whole procedure lasts approximately 15 minutes. At the end of the TSST (T1 - Post-Stress), physiological parameters via biofeedback will be measured again, and the STAI-State and SUDS questionnaires will be re-administered to assess the stress response. Immediately following this, participants will receive the intervention assigned by randomization for a duration of 30 minutes: the Experimental group will receive a diaphragmatic breathing intervention according to the Neo-Functional approach, conducted by specialized psychotherapists, involving active manual assistance to facilitate congruent respiratory movements; the Control group will rest in the same room in the presence of a therapist who, to control for the potential vagotonic effects of physical contact, will apply occasional non-specific physical contact to the participant's arm without providing breathing instructions or applying the specific diaphragmatic technique. At the end of the 30-minute intervention or control period (T2 - Post-Intervention), physiological parameters via biofeedback will be measured once more, and the STAI-State and SUDS questionnaires will be re-administered to evaluate stress recovery.

This research aims to provide initial evidence on the efficacy of a single session of Neo-Functional diaphragmatic breathing for acute stress recovery. Understanding the immediate neurobiological and psychological effects can inform the use of such techniques as accessible tools for stress management in daily life or during periods of tension. By including a control group matched for physical contact, the study aims to differentiate the specific benefits of the targeted breathing technique involving manual guidance from the more general effects of therapeutic presence and touch. The findings may contribute to the broader understanding of how targeted breathing practices influence the autonomic nervous system and subjective well-being. The psychoeducational component may also indirectly benefit participants by increasing their awareness of stress effects and potential coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aging between 18 and 55;
* Able to understanding and signing the informed consent;

Exclusion Criteria:

* a current or lifetime diagnosis of any psychiatric disorders
* a past or present of drug abuse or drug addiction (including nicotine)
* chronic inflammation diseases
* Taking medicines active on the immune system (antibiotics, anti-histamines, corticosteroids, psychotropic substances) during the 2 weeks prior to the operation;
* Intense physical activities (at least 1h\day);
* Intelligence Quotient less than 65
* BMI more than 40
* serious infections (such as HIV, hepatitis B and C)
* cancer in the previous 6 months
* regular use of anti-inflammatory drugs for more than 15 days/month
* Participation to other clinical trials;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate values | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  The difference in mean HR is an indirect measure of autonomous nervous system. It will be measured non-invasively via ProComp Infiniti photoplethysmograph. Higher values of HR represent worst parasympathetic activity.
Changes in skin conductance values | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes in mean SC values, measured non-invasively in micro-Siemens (µS) using the ProComp Infiniti physiological measurement unit. Higher SC values reflect greater physiological arousal, indicating increased sympathetic nervous system activity.
Changes in surface electromyography values on left deltoid | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes of mean EMG values, measured non-invasively in microvolts (µV) using using the ProComp Infiniti physiological measurement unit. Higher mean EMG values indicate greater muscle tension, and suggest sympathetic activation.
Changes in state anxiety | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes in state anxiety, measured by the STAI-state questionnaire. The score range from 20 to 80, with higher values indicating worst levels of anxiety.
Changes in perceived stress | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes in perceived stress measured by the SUDS questionnaire. The score ranging from 0 to 10, with higher values indicating worst levels of perceived stress.
Changes in respiratory amplitude | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes in RESP AMP were measured non-invasively using an abdominal elastic band connected to the ProComp Infiniti physiological measurement unit. The system quantifies the extent of abdominal expansion and contraction during each breath cycle, providing a measure of the depth of breathing. Higher abdominal amplitude indicate a deeper, more diaphragmatic breathing.
Changes in respiratory rate | Immediately Post-TSST (T1) and immediately post-intervention (T2)
  Changes in respiratory rate were measured using an abdominal elastic band connected to the ProComp Infiniti physiological measurement unit. The system detects the cyclical expansion and contraction of the abdomen to determine the number of BPM. A lower respiratory rate is indicative of a shift towards a more relaxed breathing pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Psychiatry of Policlinico P. Giaccone, Palermo, Italy, Italy